CLINICAL TRIAL: NCT02421159
Title: Hybrid STTR Intervention for Heterosexuals: Anonymous Testing and Confidential Care Linkage
Acronym: BCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-00963
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2017-03

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; vulnerable populations; heterosexuals at high risk; peer-driven intervention; tailored intervention; African-American; Latino/Hispanic; Seek, test, treat, and retain (STTR); Brooklyn
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Seek and Test Phase — The primary endpoint for this phase is the proportion of newly identified HIV infections of the RDS-ASTN intervention. Components for eligible and willing participants are a computerized baseline interview, counseling session, blood draw for HIV testing, HIV pre-test counseling, use of blood samples for clinical lab tests if found to be HIV infected, semi-structured interviews (if selected), the opportunity to recruit peers for the study, and the post-test counseling session.
Behavioral: Treat and Retain Phase — The primary endpoints for this phase are: proportion linked to care within three months and time to the HIV care appointment. Participants with HIV infection who are interested in participating will be enrolled in this phase and navigated to HIV primary care over three months. Components are the locator form, patient navigation and support contacts, medical report form, follow-up contacts to update locator information, semi-structured interviews, follow-up interview, and blood draw for clinical lab testing.

SUMMARY:
The Brooklyn Community United (BCU) study is a supplement to the main research study titled "Peer Driven Intervention to Seek, Test, & Treat Heterosexuals at High Risk for HIV." The main study's field name is Brooklyn Community Action Project (BCAP) (R01DA032083, R#: 11-01257). The main study is testing two approaches to seeking out undiagnosed HIV infection (Venue-based Sampling (VBS) and Confidential Two-Session Testing with Navigation (CTTN-RDS)).

HIV prevalence rates in two previous heterosexual cycles of NHBS in the local area are: 7% in HET1 and 12.3% in HET2. The main study, BCAP, found lower prevalence rates of 3.45%, 35.14% of which were newly diagnosed in the RDS-CTTN sample and 1.89% newly diagnosed with HIV in the VBS sample.

The primary aim of the Brooklyn Community United (BCU) study is to seek out individuals with undiagnosed HIV using a streamlined RDS-CTTN approach, and anonymous HIV Testing in Central Brooklyn.

The supplement study hypotheses are:

(H1): Compared with VBS and RDS-CTTN, and controlling for potential differences on key socio-demographic characteristics across the samples, RDS-ASTN participants will have less HIV testing experience.

(H2) Controlling for potential differences on key socio-demographic characteristics across the samples, RDS-ASTN will yield higher rates previously undiagnosed HIV compared with VBS and RDS-CTTN.

(H3): Most participants (> 70%) found to be HIV-infected in the RDS-ASTN intervention will engage in the Treat and Retain intervention phase.

(H4): Most participants in the Treat and Retain phase of the RDS-ASTN intervention (> 70%), all of whom will be HIV infected, will be linked to care within 3 months.

DETAILED DESCRIPTION:
The Brooklyn Community United (BCU) study is a supplement to the main research study to seek, test, treat and retain heterosexuals at high risk for HIV. The main research study is entitled "Peer Driven Intervention to Seek, Test, & Treat Heterosexuals at High Risk for HIV." The main study's field name is Brooklyn Community Action Project or BCAP (R01DA032083, R#: 11-01257). The main study is testing two approaches to seeking out undiagnosed HIV infection (Venue-based Sampling and Confidential Two-Session Testing with Navigation).

We have studied HHR in New York City as part of the CDC's National HIV Behavioral Surveillance (NHBS) studies. Building on the NHBS work, we are currently in our third year of the main study (R01DA032083, R#: 11-01257), the primary aim of which is to compare the efficacy of a peer-driven intervention that uses a respondent-driven sampling strategy ("RDS-CTTN") and venue-based sampling (VBS) with respect to identifying previously undiagnosed HIV infection. The main study is located in central Brooklyn, a high-risk area (HRA) with elevated rates of poverty, high heterosexual HIV prevalence, and where a generalized HIV epidemic may be said to exist.

To date, RDS-CTTN and VBS have enrolled approximately 45% of their samples (RDS-CTTN 1338/3000; VBS 174/400). Participants in both samples evidence high rates of risk factors (substance use, incarceration, homelessness, unemployment). As hypothesized, PDI/RDS is reaching a population with higher rates of risk factors, and lower rates of HIV testing compared to VBS. Almost all in RDS-CTTN and VBS had been tested at least once previously (> 86%), but fewer than half have been tested in the past year. Among those with lifetime testing, data suggest testing is infrequent with a median of 2.5 tests per ten years of adulthood. Interestingly, almost all of those who enroll in RDS-CTTN and VBS elected to test for HIV (> 90%), with no difference in HIV testing acceptance rates between those who tested previously and first-time testers. This suggests that those who enroll in the study, although they have known barriers to HIV testing and a range of risk factors for adverse outcomes, are open to confidential HIV testing. These findings support the promise of the RDS-CTTN approach, but preliminary studies also signal the need to reach those with the greatest fears of and barriers to HIV testing who will not engage in confidential testing.

With approximately 45% of the sample enrolled, HIV prevalence in the RDS-CTTN sample is 3.45% (37/1071); 35.14% of these are newly diagnosed (13/37). Rates of newly diagnosed HIV infection may continue to increase as recruitment chains reach deeper into hidden and more vulnerable components of networks. In VBS, 1.89% is newly diagnosed with HIV (3/159). Yet these HIV prevalence rates are lower than those found in two previous heterosexual cycles of NHBS in the local area: 7% in HET1 and 12.3% in HET2 spurring our interest in additional innovative strategies to seek out those with undiagnosed HIV.

Despite its high acceptability among enrolled participants and preliminary evidence of efficacy, the two-session RDS-CTTN approach may be less successful in enrolling those in the HRA who would decline confidential HIV testing in a formal setting or have poor access to such testing. The RDS-CTTN intervention may not be optimal for reaching those with the greatest psychosocial barriers to regular HIV testing, who may for a number of reasons have high rates of undiagnosed HIV, or individuals, particularly women, with multiple job and family responsibilities who may not have time for a two-session intervention. (Indeed women are under-represented in both RDS-CTTN [~ 40%] and VBS [~30%].) It is possible to test participants for HIV in a first encounter, aswe do in VBS and as other studies have done. In the supplement study, we build on lessons learned from themain study in progress and the literature to address this concern.

Anonymous testing is available in state and local health departments, in cases of occupational exposure, through home test/self-test technologies, and research studies including our local NHBS studies with HHR. There is some evidence to suggest individuals who test anonymously do so earlier in the course of their HIV disease than those who engage in confidential testing. Additionally, anonymous testing may be useful for and/or preferred by individuals from marginalized populations. As Kegeles and colleagues have found, many who seek anonymous HIV-antibody testing would avoid it under other circumstances, and anonymous testing may be preferred among those who suspect they are infected, and by bisexual individuals, and those who fear stigma and discrimination. Thus, a brief, anonymous HIV testing effort may appeal to and engage HHR who face barriers to confidential HIV testing.

While anonymous testing may be an effective and/or efficient strategy in the 'seek' phase of STTR, in the majority of studies and testing programs it does not address the vital step of linkage to care. Although anonymous testing tends to yield individuals earlier in their HIV disease, those who test anonymously are more likely to experience delays entering care, because anonymous testing sites and programs do not typically have the resources to engage individuals into linkage programs and are not co-located with medical care. For example, in a study of characteristics of the HIV testing encounter and linkage to care, Reed (2009) found that 36% of those testing anonymously did not enter care within three months of diagnosis, compared with 26% of those testing confidentially.

The supplement study hypotheses are:

(H1): Compared with VBS and RDS-CTTN, and controlling for potential differences on key socio-demographic characteristics across the samples, RDS-ASTN participants will have less HIV testing experience.

(H2) Controlling for potential differences on key socio-demographic characteristics across the samples, RDS-ASTN will yield higher rates previously undiagnosed HIV compared with VBS and RDS-CTTN.

(H3): Most participants (> 70%) found to be HIV-infected in the RDS-ASTN intervention will engage in the Treat and Retain intervention phase.

(H4): Most participants in the Treat and Retain phase of the RDS-ASTN intervention (> 70%), all of whom will be HIV infected, will be linked to care within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* sexually active (vaginal, anal) with at least one partner of the opposite sex within the previous year;
* reside in the 7 zip code central Brooklyn HRA (initial seeds only; peers may reside in the larger 19 zip code HRA);
* comprehend English or Spanish;
* HIV negative or unknown HIV status (initial seeds only; peers may be 'known positives');
* willing to try to recruit peers;

Exclusion Criteria:

* actively psychotic based on valid screening instrument;
* participant in the past NHBS studies with HHR (called HET1, 2, 3);
* enrolled already in the supplement study (RDS-ASTN), VBS or RDS-CTTN in the main study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
proportion of newly diagnosed HIV infections | 1 week post-baseline

SECONDARY OUTCOMES:
proportion linked to care | 3 months post-baseline
time to the HIV care appointment | 3 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marya Gwadz, PhD, Principal Investigator — New York University
Locations (1):
- New York University College of Nursing, New York, New York, United States

REFERENCES:
- [Derived] Gwadz M, Cleland CM, Leonard NR, Kutnick A, Ritchie AS, Banfield A, Hagan H, Perlman DC, McCright-Gill T, Sherpa D, Martinez BY; BCAP Collaborative Research Team. Hybrid STTR intervention for heterosexuals using anonymous HIV testing and confidential linkage to care: a single arm exploratory trial using respondent-driven sampling. BMC Public Health. 2015 Nov 16;15:1133. doi: 10.1186/s12889-015-2451-5. PMID 26572865